CLINICAL TRIAL: NCT00519064
Title: A Phase III, Randomized, Controlled, Observer-blind, Single-center Study to Compare Immunogenicity and Safety of an Adjuvanted Inactivated Subunit Influenza Vaccine to Those of a Non-adjuvanted Inactivated Subunit Influenza Vaccine, When Administered to Adults Affected by Chronic Diseases
Brief Title: Immunogenicity and Safety of an Adjuvanted Inactivated Subunit Influenza Vaccine to Those of a Non-adjuvanted Inactivated Subunit Influenza Vaccine, When Administered to Adults Affected by Chronic Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V70P3; 2006-005558-63
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-02

CONDITIONS: Influenza Disease
Keywords: influenza; influenza vaccine; adjuvanted influenza vaccine; H5N1 influenza antigen
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Biological: Adjuvanted influenza vaccine
- Arm 2 (Active Comparator)
  Interventions: Biological: Adjuvanted influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted influenza vaccine

SUMMARY:
This phase III is designed to confirm the previous trial results evaluating the safety, clinical tolerability and immunogenicity of the 2006-2007 formulation of Novartis Vaccines' adjuvanted influenza vaccine and subunit influenza vaccine in adults with underlying chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years of age adult volunteers, mentally competent, willing and able to give written informed consent prior to study entry, suffering from at least one of these chronic diseases:moderate to severe hypertension, moderate to severe congestive heart failure, chronic obstructive pulmonary disease (COPD) or moderate to severe asthma, moderate to severe hepatic or renal insufficiency, arteriosclerotic disease or insulin dependent diabetes mellitus

Exclusion Criteria:

* Hypersensitivity to ovalbumin, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine;
* History of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine;
* Known or suspected impairment/ alteration of immune function;
* Any condition which might interfere with the evaluation of the study objectives

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 361 (Actual)
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Compare immunogenicity of a single IM inj. of an adj. inactivated subunit flu vaccine vs. inactivated subunit virus flu vaccine, with regards to A/H3N2 antigen, when administered to adults with underlying chronic disease, as measured by HI test at day 22

SECONDARY OUTCOMES:
Compare immunogenicity of an IM injection of an adj. inactivated subunit flu vaccine vs. inactivated subunit virus flu vaccine, with regards to B antigen, when administered to adults with underlying chronic disease, as measured by HI test at day 22
Evaluate immunog. of a single IM inj. of an adj. inactivated subunit flu vaccine vs. inactivated subunit virus flu vaccine, with regards to A/H1N1 antigen, when administered to adults with underlying chronic disease, as measured by HI test at day 22
To evaluate the safety of a single IM injection of the two influenza vaccines, when administered to adult subjects with underlying chronic disease(s).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- Azienda ULSS 13 di Mirano, Mira, Via Nazionale 48, Venezia, Italy

REFERENCES:
- [Result] Black S, Della Cioppa G, Malfroot A, Nacci P, Nicolay U, Pellegrini M, Sokal E, Vertruyen A. Safety of MF59-adjuvanted versus non-adjuvanted influenza vaccines in children and adolescents: an integrated analysis. Vaccine. 2010 Oct 21;28(45):7331-6. doi: 10.1016/j.vaccine.2010.08.075. Epub 2010 Sep 15. PMID 20813217